CLINICAL TRIAL: NCT01999660
Title: Prospective National Post-marketing Surveillance for the Investigation of the Efficacy and Safety of SpaceOAR™ to Maintain Space Between the Rectum and Prostate During Radiation Therapy
Brief Title: Post-marketing Surveillance Regarding Efficacy and Safety of SpaceOAR™
Status: Terminated | Type: Observational
Why Stopped: PI did leave hospital (retired)
Sponsor: CS Diagnostics GmbH (Industry)
Collaborators: Aix Scientifics (Industry)
Responsible Party: Sponsor
Other Study IDs: Space-CS-01
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer Patients Treated by Radiotherapy
Keywords: Prostatic Neoplasms; Radiotherapy; rectal toxicity
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SpaceOAR™: prostate cancer patient prophetically treated by SpaceOAR™
  Interventions: Device: SpaceOAR™ implantation

INTERVENTIONS:
Device: SpaceOAR™ implantation

SUMMARY:
A treatment with SpaceOAR™ hydrogel does reduce late toxicity Grad 2 and Grad 3 of radiation therapy in prostate cancer patients

DETAILED DESCRIPTION:
The degradable SpaceOAR™ hydrogel establishes for the time of radiotherapy a distance between the prostate and the rectum

ELIGIBILITY:
Inclusion Criteria:

* Patient is suffering from pathologically confirmed T1-T2, N0, M0 prostate adenocarcinoma.
* Patient is intended to receive radiation therapy (3D-computerized radiotherapy, intensity-modulated radiotherapy, and/or brachytherapy) and this will be the first prostate or pelvic radiation therapy.
* Patient is intended to receive SpaceOAR™ Gel therapy.
* The patient is official patient of the clinical investigator in the study centre.
* Patient agrees to fully participate in the clinical trial and give informed consent in writing.

Exclusion Criteria:

* Anatomic abnormality, physical or pathological condition precluding the implantation.
* Failure in the wall of the perineum room (with the risk that the hydrogel escapes).
* History of prostate surgery or local prostate cancer therapy.
* Rectal injury before implantation of SpaceOAR™ Gel or history of or active inflammatory rectal disease such as Crohn's disease or ulcerative colitis.
* History of or current perirectal or anal disease or surgery such as prolapsed or bleeding haemorrhoids or fistula.
* Compromised immune system (e.g., HIV/acquired immunodeficiency syndrome, auto¬immune disease or immunosuppressive therapy).
* Platelet count, partial thromboplastin time, or white blood cell count out of normal laboratory range.
* Contraindication for safe MRI and CT scans.
* Patient is not able to fully participate in this study including the follow-up (e.g. for mental or geographical reasons, or patient is intravenous drug user or has strong potential for non-compliance to medical regimes).
* Patient is mentally unable to understand the nature, aims, or possible consequences of the clinical investigation.
* Patient has restricted legal capacity.
* Patient did participate in another clinical investigation during the last 3 months.
* Patient has revoked the consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prostate cancer patients treated by radiotherapy and prophetically by SpaceOAR™
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2013-11; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
the rectal complication rate (late toxicity) | 6 months and yearly for 5 years thereafter
  the rectal complication rate following the common toxicity criteria (CTC) v. 2.0

SECONDARY OUTCOMES:
Quality of Life | 6 months and for 5 years yearly thereafter
  The validated Expanded Prostate Cancer Index Composite (EPIC) questionnaire in combination with the validated Short Form Health Survey (SF-12) will be used to document the influence on the quality of life (QoL).

OTHER OUTCOMES:
feasibility of the implantation procedure | 1 day
  feasibility of the implantation procedure will be documented by subjective description given by the investigators. this includes safety aspects.

CONTACTS AND LOCATIONS:
Overall Officials: Razvan Galalae, PD Dr. med., Principal Investigator — Clinic for Radiooncology and Radiotherapy, Evangelical Clinics Gelsenkirchen, Germany
Locations (1):
- Clinic for Radiooncology and Radiotherapy, Evangelical Clinics Gelsenkirchen, Gelsenkirchen, North Rhine-Westphalia, Germany